CLINICAL TRIAL: NCT03117569
Title: A Phase IIIb, Open-label, Multicentre, International Randomised Controlled Trial of Simplified Treatment Monitoring for 8 Weeks Glecaprevir (300mg)/Pibrentasvir (120mg) in Chronic HCV Treatment naïve Patients Without Cirrhosis
Brief Title: Trial of Simplified Treatment Monitoring for 8 Weeks Glecaprevir/Pibrentasvir in Chronic Hepatitis C Patients
Acronym: SMART-C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VHCRP1701
Record Dates: First submitted 2017-04-07; First posted 2017-04-18 (Actual); Results first posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — glecaprevir; pibrentasvir; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard monitoring schedule (Other): Participants will have on-treatment clinic visits at weeks 4 and 8. Participants have also phone contact-based visits at weeks 4 and 8 (1-2 days prior to scheduled clinic visits).
  Interventions: Drug: glecaprevir (300mg)/pibrentasvir (120mg)
- Simplified monitoring schedule (Experimental): Participants will have no on-treatment clinic visits at weeks 4 and 8. Participants have phone contact-based visits at weeks 4 and 8.
  Interventions: Drug: glecaprevir (300mg)/pibrentasvir (120mg)

INTERVENTIONS:
Drug: glecaprevir (300mg)/pibrentasvir (120mg) — glecaprevir (300mg)/pibrentasvir (120mg) for 8 weeks
  Other Names: Mavyret

SUMMARY:
The aim of this study is to determine if treatment monitoring schedule for chronic HCV patients treated with glecaprevir (300mg)/pibrentasvir (120mg) can be simplified.

Data has shown that direct acting antiviral (DAA) regimen of glecaprevir (300mg)/pibrentasvir (120mg), a protease inhibitor and NS5A inhibitor respectively , provides key features for HCV treatment simplification.

Eligible participants (naïve pre-cirrhosis chronic HCV patients) will be randomized (1:2) to the standard or simplified monitoring arm and will receive treatment for 8 weeks.

One post treatment visit will be conducted 12 weeks after the final dose of study medication to evaluate the proportion of patients with undetectable HCV RNA at this timepoint (SVR12).

DETAILED DESCRIPTION:
The capacity to scale-up interferon-free DAA therapy would be enhanced by simplified treatment monitoring strategies. The "next generation" DAA regimen of glecaprevir (300mg)/pibrentasvir (120mg), a protease inhibitor and NS5A inhibitor, provides key features for HCV treatment simplification, including on-treatment monitoring: 1) pangenotypic activity with extremely high efficacy (SVR>95%); 2) no relationship between time to undetectable HCV RNA and SVR; 3) minimal drug-related toxicity; 4) ease of dosing (three pills once daily); and short duration (8 weeks in non-cirrhosis and 12 weeks in cirrhosis for treatment naïve patients). In phase II and III clinical trials in participants without cirrhosis, 8 weeks of glecaprevir (300mg)/pibrentasvir (120mg) has provided intention-to-treat SVR rates of 99.1%, 98%, 97%, and 93.1% in genotype 1, 2, 3, and 4-6 populations, respectively.

Current standard on-treatment monitoring in clinical trials involves clinic-based visits every 4 weeks. In the DAA era where treatments are highly tolerable, effective and short duration, this intensive monitoring strategy may no longer be required. A simplified on-treatment monitoring strategy is hypothesised to be non-inferior to the standard clinical trial on treatment monitoring strategy. If successful, a simplified on-treatment monitoring strategy is likely to be highly attractive to patients, clinicians and health care payers. It has the potential to improve the rapid scale up of treatment providing population level benefits in the reduction of global hepatitis C disease burden.

This study will be conducted as a Phase IIIb, randomised, controlled, multicentre, international trial.

There will be a maximum screening period of 6 weeks prior to Baseline. Eligible patients will be randomised into one of two on-treatment monitoring strategies; standard clinical trial monitoring (4-weekly on-treatment visits) vs simplified monitoring (no on-treatment visits). Randomisation will be 1:2 (standard vs simplified) and all participants will receive treatment with glecaprevir (300mg)/pibrentasvir (120mg) for 8 weeks.

All participants will attend the clinic for screening and baseline visit. Randomisation will occur at the baseline visit.

The two on-treatment monitoring strategies will differ as follows:

* Standard monitoring arm participants will have on-treatment clinic visits at weeks 4 and 8 (EoT).
* Simplified monitoring arm participants will have no on-treatment clinic visits.

Study nurse phone contact will also be made to participants in BOTH arms 1-2 days prior Week 4 and EoT (Week 8) visits to provide standardized reporting of adverse events, concomitant medication and adherence. One post treatment clinic visit will be conducted at SVR12 (week 20) for all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Have voluntarily signed the informed consent form.
2. 18 years of age or older.
3. Chronic HCV infection as defined by anti-HCV antibody or HCV RNA detection for greater than 6 months.
4. HCV RNA plasma ≥ 10,000 IU/ml at screening.
5. HCV genotype 1-6.
6. HCV treatment naïve (no prior treatment with an approved or investigation anti-HCV medication).
7. Stage F0-3, based on: hepatic elastography <12.5 kPa on Fibroscan® or APRI <1.0.
8. If co-infection with HIV is documented, the subject must meet the following criteria:

   * ART naïve with CD4 T cell count >500 cells/mm3; OR
   * On a stable ART regimen (containing only permissible ART - see protocol section 3.2) for >8 weeks prior to screening visit, with CD4 T cell count >200 cells/mm3 and a plasma HIV RNA level below the limit of detection.
9. Negative pregnancy test at screening and baseline (females of childbearing potential only).
10. All fertile females must be using effective contraception during treatment and during the 30 days after treatment end.

Exclusion Criteria:

1. History of any of the following:

   1. Clinically significant illness (other than HCV) or any other major medical disorder that may interfere with the participant treatment, assessment or compliance with the protocol; participants currently under evaluation for a potentially clinically significant illness (other than HCV) are also excluded.
   2. Clinical hepatic decompensation (i.e. ascites, encephalopathy or variceal haemorrhage).
   3. Solid organ transplant.
   4. History of severe, life-threatening or other significant sensitivity to any excipients of the study drugs.
2. Any of the following lab parameters at screening:

   1. ALT > 10 x ULN
   2. AST > 10 x ULN
   3. Direct bilirubin > ULN
   4. Platelets < 90,000/μL (cells/mm3) if Fibroscan® <12.5 kPa OR < 150,000/μL (cells/mm3) if Fibroscan® is unavailable and patient is included with APRI <1
   5. Creatinine clearance (CLcr) < 50 mL/min
   6. Haemoglobin < 12g/dL for males; <11g/dL for females
   7. Albumin < LLN
   8. INR > 1.5 ULN unless subject has known haemophilia or is stable on an anticoagulant regimen affecting INR
3. Pregnant or breastfeeding female.
4. HBV infection (HBsAg positive).
5. Use of prohibited concomitant medications as described in protocol section 5.2.
6. Chronic use of systemically administered immunosuppressive agents (e.g. prednisone equivalent > 10 mg/day for >2 weeks).
7. Therapy with any anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) ≤6 months prior to the first dose of study drug.
8. Any investigational drug ≤6 weeks prior to the first dose of study drug.
9. Ongoing severe psychiatric disease as judged by the treating physician.
10. Positive result of a urine drug screen at the Screening Visit for opiates, barbiturates, amphetamines, cocaine, benzodiazepines, phencyclidine, propoxyphene, or alcohol, with the exception of a positive result (including methadone) associated with documented short-term use or chronic stable use of a prescribed medication in that class.
11. Injecting drug use within the previous six months.
12. Inability or unwillingness to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Dore, Principal Investigator — Kirby Institute, University of New South Wales Sydney, Australia
Locations (33):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - New York University Langone Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - SSM Health Dean Medical Group, Madison, Wisconsin
- Australia (6):
  - East Sydney Doctors, Sydney, New South Wales
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - St Vincent's Hospital Melbourne, Melbourne, Victoria
- Canada (7):
  - Lair Centre, Vancouver, British Columbia
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - William Osler Health System, Brampton, Ontario
  - St Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
- France (3):
  - Hopital Henri Mondor, Créteil
  - Hopital Saint Joseph, Marseille
  - Hopital Saint Antoine, Paris
- Germany (4):
  - zibp - Zentrum für Infektiologie Berlin Prenzlauer Berg GmbH, Berlin
  - Center for HIV and Hepatogastroenterology, Düsseldorf
  - Hannover Medical School, Hanover
  - CIM-Centrum fuer Interdisziplinaere Medizin GmbH, Münster
- New Zealand (4):
  - Auckland City Hospital, Auckland
  - Calder Center, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern, Bern
  - University Hospital Zurich, Zurich
- United Kingdom (3):
  - Barts Health, London
  - King's College Hospital, London
  - Imperial College Healthcare NHS Trust (St Mary's Hospital), London

IPD SHARING:
Plan to Share IPD: Yes
No individual participant data will be shared. The results of the project will be presented at scientific meetings, and published in peer reviewed scientific literature. Sharing of data generated by this project is an essential part of our proposed activities and will be carried out in several different ways. We plan to make our results available to the community of scientists interested in recently acquired hepatitis C, community organisations representing the affected communities and participants. We also welcome collaboration with others who could make use of data and samples.
Supporting Information: Study Protocol, SAP
Time Frame: Submitted as part of J Hepatology accepted publication
Access Criteria: Access via the J Hepatology accepted publication

REFERENCES:
- [Derived] Dore GJ, Feld JJ, Thompson A, Martinello M, Muir AJ, Agarwal K, Mullhaupt B, Wedemeyer H, Lacombe K, Matthews GV, Schultz M, Klein M, Hezode C, Mercade GE, Kho D, Petoumenos K, Marks P, Tatsch F, Dos Santos AGP, Gane E; SMART-C Study Group. Simplified monitoring for hepatitis C virus treatment with glecaprevir plus pibrentasvir, a randomised non-inferiority trial. J Hepatol. 2020 Mar;72(3):431-440. doi: 10.1016/j.jhep.2019.10.010. Epub 2019 Oct 23. PMID 31655134

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 21 August 2017 to 16 July 2018, participants were screened and enrolled at 33 sites in Australia (n=6), Canada (n=7), France (n=3), Germany (n=4), New Zealand (n=4), Switzerland (n=2), United Kingdom (n=3), and United States (n=4). Study recruitment was in tertiary specialist viral hepatitis clinics (n=30) and primary care clinics (n=3).
Groups:
- Standard Monitoring Schedule: Participants will have on-treatment clinic visits at weeks 4 and 8. Participants have also phone contact-based visits at weeks 4 and 8 (1-2 days prior to scheduled clinic visits).
  Participants receive glecaprevir (300mg)/pibrentasvir (120mg): glecaprevir (300mg)/pibrentasvir (120mg) for 8 weeks
- Simplified Monitoring Schedule: Participants will have no on-treatment clinic visits at weeks 4 and 8. Participants have phone contact-based visits at weeks 4 and 8.
  Participants receive glecaprevir (300mg)/pibrentasvir (120mg): glecaprevir (300mg)/pibrentasvir (120mg) for 8 weeks
Period: Overall Study
Arm/Group | Standard Monitoring Schedule | Simplified Monitoring Schedule
Started | 127 | 253
Completed | 123 | 241
Not Completed | 4 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Monitoring Schedule | Simplified Monitoring Schedule | Total
Number analyzed (Participants) | 127 | 253 | 380
Age, Continuous [Mean (Full Range); unit: Years] | 50 [24 to 79] | 52 [22 to 73] | 51 [22 to 79]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 72 | 157 | 229
  Gender: Female | 53 | 96 | 149
  Gender: Transgender | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 97 | 194 | 291
  Ethnicity: Asian | 12 | 22 | 34
  Ethnicity: Black | 7 | 13 | 20
  Ethnicity: Other | 11 | 24 | 35
Region of Enrollment [Number; unit: participants]
  New Zealand | 29 | 57 | 86
  Canada | 28 | 58 | 86
  United States | 11 | 22 | 33
  United Kingdom | 9 | 15 | 24
  Australia | 15 | 30 | 45
  France | 14 | 28 | 42
  Switzerland | 8 | 15 | 23
  Germany | 13 | 28 | 41
HCV RNA [Median (Full Range); unit: Log10 IU/mL] | 6.29 [2.85 to 7.71] | 6.27 [2.49 to 7.74] | 6.28 [2.49 to 7.74]
Genotype [Count of Participants; unit: Participants]
  Genotype 1 | 61 | 118 | 179
  Genotype 2 | 17 | 35 | 52
  Genotype 3 | 41 | 80 | 121
  Genotype 4 | 4 | 14 | 18
  Genotype 5 | 1 | 0 | 1
  Genotype 6 | 3 | 5 | 8
  Indeterminate | 0 | 1 | 1
Fibrosis Stage [Count of Participants; unit: Participants]
  No or mild fibrosis (F0/F1) | 93 | 190 | 283
  Mild fibrosis (F2) | 29 | 49 | 78
  Severe fibrosis (F3) | 5 | 14 | 19
HIV Infection [Count of Participants; unit: Participants] | 13 | 14 | 27
Opioid Substitution Therapy (OST) [Count of Participants; unit: Participants] | 17 | 21 | 38

OUTCOME MEASURES:

1. Primary Outcome: Undetectable HCV RNA (ITT Population)
Description: Number of participants with undetectable HCV RNA based on ITT population.
Time Frame: 12 weeks post end of treatment (SVR12)
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Monitoring Schedule | Simplified Monitoring Schedule
Number analyzed (Participants) | 127 | 253
Participants | 121 | 233
Statistical Analysis 1: Comparison: Standard Monitoring Schedule vs Simplified Monitoring Schedule; Test type: Non-Inferiority — A total of 375 participants (2:1 randomisation) were planned for enrolment and evaluation as ITT population. Under the assumption that SVR12 rate would be 96% in both arms, the study had 80% power to show non-inferiority of the simplified monitoring strategy with a lower confidence bound for SVR12 in the simplified monitoring arm greater than 90% or with a lower confidence bound for the difference (simplified arm minus standard arm) in SVR12 greater than -6%; p < 0.05, t-test, 2 sided; Difference in Percentage of Participants = -3.2, 95% CI 2-sided [-8.2 to 1.8]

2. Secondary Outcome: Undetectable HCV RNA (mITT Population)
Description: Number of participants with undetectable HCV RNA based on mITT population.
Time Frame: 12 weeks post end of treatment (SVR12)
Population: The mITT population wexcludes patients who have completed treatment (>95% adherence) (according to phone contact at week 8), but have not returned for their SVR12 assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Monitoring Schedule | Simplified Monitoring Schedule
Number analyzed (Participants) | 123 | 241
Participants | 121 | 233

3. Secondary Outcome: Treatment and Study Visits Adherence
Description: Number adherent to treatment and study visits (on-treatment adherence and early treatment discontinuation).
Time Frame: 12 weeks post end of treatment (SVR12)
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Monitoring Schedule | Simplified Monitoring Schedule
Number analyzed (Participants) | 127 | 253
Participants
  >=95% Adherence | 125 | 241
  <95% Adherence | 2 | 12

4. Secondary Outcome: Health-related Quality of Life
Description: Change in health-related quality of life score pre and post-treatment (measured by EQ-5D-3L). The EQ visual analogue scale records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' (value of 100) and 'Worst imaginable health state' (value of 0). The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement. Higher scores indicate better outcomes.
Time Frame: Screening and 12 weeks post end of treatment (SVR12)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard Monitoring Schedule | Simplified Monitoring Schedule
Number analyzed (Participants) | 127 | 253
score on a scale
  Screening | 80 [20 to 100] | 80 [40 to 100]
  Post-treatment week 12 | 85 [20 to 100] | 89 [40 to 100]

5. Secondary Outcome: Number of Virological Failure Participants With NS3 and NS5A Polymorphisms at Baseline and Post-treatment Week 12
Description: Distribution of baseline resistance associated substitutions (RAS) in participants with virological failures. Baseline polymorphisms were detected by Sanger sequencing at the following amino acid positions:
  NS3: 36, 56, 80, 155, 156, 166, 168 NS5A: 24, 28, 30, 31, 58, 93
Time Frame: Baseline and 12 weeks post-treatment
Population: Number of participants in the ITT population with virological failure (detectable HCV RNA)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Monitoring Schedule | Simplified Monitoring Schedule
Number analyzed (Participants) | 2 | 6
Participants
  NS3 Variants at Baseline | 0 | 1
  NS3 Variants at Failure | 1 | 3
  NS5A Variants at Baseline | 0 | 3
  NS5A Variants at Failure | 0 | 5

6. Secondary Outcome: Patient Treatment Satisfaction
Description: Patient was satisfied with their treatment follow-up plan.
Time Frame: 12 weeks post end of treatment (SVR12)
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Monitoring Schedule | Simplified Monitoring Schedule
Number analyzed (Participants) | 127 | 253
Participants
  Strongly Disagree | 1 | 4
  Disagree | 0 | 2
  No Opinion | 3 | 9
  Agree | 29 | 61
  Strongly Agree | 83 | 149
  Missing | 11 | 28

7. Other Pre Specified Outcome: Common Adverse Events (Safety Outcome)
Description: Proportion of patients with common adverse events (reported in greater than 5%).
Time Frame: 12 weeks post end of treatment (SVR12)
Population: ITT
Measure: Number; unit: participants
Arm/Group | Standard Monitoring Schedule | Simplified Monitoring Schedule
Number analyzed (Participants) | 127 | 253
participants
  Fatigue | 30 | 52
  Headache | 26 | 43
  Nausea | 25 | 17

8. Other Pre Specified Outcome: Severe/Life Threatening Adverse Events (Safety Outcome)
Description: Proportion of patients with at least one severe or potentially life threatening (grade 3 or 4) adverse event.
Time Frame: 12 weeks post end of treatment (SVR12)
Population: ITT
Measure: Number; unit: participants
Arm/Group | Standard Monitoring Schedule | Simplified Monitoring Schedule
Number analyzed (Participants) | 127 | 253
participants | 1 | 2

9. Other Pre Specified Outcome: Provider Acceptability of Simplified Monitoring Strategy (Exploratory Outcome)
Description: Provider acceptability of simplified monitoring strategy measured by study specific questionnaire completed by each site Principal Investigator and the primary Research Nurse.
Time Frame: 12 weeks post end of treatment (SVR12)
Measure: Count of Participants; unit: Participants
Groups:
- Screening: Health Practitioner attitudes regarding the model of care as expressed via questionnaire completed prior to first patient first visit.
- Post Treatment Week 12: Health Practitioner attitudes regarding the model of care as expressed via questionnaire completed after the last patient last visit.
Arm/Group | Screening | Post Treatment Week 12
Number analyzed (Participants) | 66 | 62
Participants
  Prefers Standard Monitoring | 14 | 7
  Prefers Simplified Monitoring | 52 | 54
  Other | 0 | 1

ADVERSE EVENTS:
Time Frame: Any treatment emergent adverse events up to 30 days after last dose
Arm/Group | Standard Monitoring Schedule | Simplified Monitoring Schedule
All-Cause Mortality (participants affected / at risk) | 0/127 | 1/253
Serious Adverse Events (participants affected / at risk) | 0/127 | 3/253
Other Adverse Events (participants affected / at risk) | 81/127 | 112/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Monitoring Schedule (N=127) | Simplified Monitoring Schedule (N=253)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Lung adenocarcinoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Monitoring Schedule (N=127) | Simplified Monitoring Schedule (N=253)
Fatigue (General disorders) | 30 | 52
Headache (Nervous system disorders) | 26 | 43
Nausea (Gastrointestinal disorders) | 25 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT03117569/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT03117569/SAP_001.pdf